CLINICAL TRIAL: NCT03529253
Title: Effect of Alirocumab(Proprotein Convertase Subtilisin/Kexin type9 Inhibitor) and Rosuvastatin or Rosuvastatin Alone on Lipid Core Plaques in Coronary Artery Disease Evaluated by Near-infrared Spectroscopy Intravascular Ultrasound
Acronym: ANTARES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, senior lecturer, Kobe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 290068
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Alirocumab; NIRS-IVUS; LCBI
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive therapy group (Experimental): Alirocumab group is Alirocumab75mg/2week plus Rosuvastatin10mg/daily.
  Interventions: Drug: Alirocumab 75 MG/ML [Praluent]+ Rosuvastatin 10mg/daily
- Standard therapy group (Active Comparator): The standard therapy group is Rosuvastatin10mg/daily alone.
  Interventions: Drug: Rosuvastatin calcium10mg

INTERVENTIONS:
Drug: Alirocumab 75 MG/ML [Praluent]+ Rosuvastatin 10mg/daily — Alirocumab group receive Alirocumab75mg/2week subcutaneous injection plus Rosuvastatin10mg/daily by oral for 9 months.
  Arms: Intensive therapy group
Drug: Rosuvastatin calcium10mg — Rosuvastatin10mg/daily by oral for 9 months.
  Arms: Standard therapy group

SUMMARY:
The purpose of this study is to verify whether additional administration of Alirocumab exerts a stronger stabilizing effect on the vulnerable plaque in CAD, compared with statin alone administration in patients receiving PCI. Therefore, the change in maxLCBI (4 mm) of the coronary artery 9 months after administration by addition administration of Alirocumab is evaluated as the main evaluation item as compared with statin administration alone for patients who have CAD and received PCI. Also, change of plaque properties is compared with baseline and evaluated. This study is a single-center, randomized, open-label study, using alirocumab, rosuvastatin as test drugs. Based on the findings obtained in this study, it is possible to clarify the mechanism of stabilization of the plaque in a patient with coronary artery disease, which in turn suppresses the progress of plaque in coronary artery disease, resulting in primary or secondary There is a possibility that it can contribute to prevention.

DETAILED DESCRIPTION:
The investigators investigate the change in the maxLCBI (4 mm) value calculated by NIRS-IVUS at the time of PCI and at the treatment evaluation after 9 months compared with the group of Alirocumab(Alirocumab75mg/2week+losuvastatin10mg/daily) and standard treatment (losuvastatin10mg/daily alone). And also the investigators evaluate LCBI(lesion), Angle of a lipid core, EEM CSA, Lumen CSA, Minimum lumen diameter, Plaque burden, Lesion length by NIRS-IVUS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent PCI for ACS or stable coronary heart disease
* Patients with LDL-C ≥70 mg/dL under daily 10mg rosuvastatin
* Patients who remained 25-75% stenosis with coronary angiography
* Patients who obtained analyzable images and calculated maxLCBI (4 mm) with NIRS-IVUS
* Patients aged ≥20 years old at PCI
* Patients who agree to be enrolled in the trial give signed written informed consent

Exclusion Criteria:

* Patients who have been treated previously with at least one dose of any anti-PCSK9 monoclonal antibody
* Patients had uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) between the time of PCI and randomization visit
* Known hypersensitivity to alirocumab or rosuvastatin
* All contraindications to alirocumab and/or rosuvastatin as displayed in the respective national product labeling for these treatments
* Known history of hemorrhagic stroke
* Currently under treatment for cancer
* Patients on lipoprotein apheresis
* Patients with severe liver or renal dysfunction
* Pregnant or breastfeeding women
* Patients recognized as inadequate by attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
maxLCBI (4mm) | baseline and 9 months

SECONDARY OUTCOMES:
change amount of LCBI(lesion) | baseline and 9 months
change amount of Angle of lipid core | baseline and 9 months
change amount of LDL-Cholesterol level | baseline and 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Undecided